CLINICAL TRIAL: NCT04653558
Title: Clinical Manifestations and Long-Term Outcome in Early Lyme Neuroborreliosis According to Diagnostic Certainty
Brief Title: Clinical Manifestations and Long-Term Outcome in Early Lyme Neuroborreliosis
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Daša Stupica, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: LNB-2020
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Lyme Disease
Keywords: Lyme neuroborreliosis; post-Lyme borreliosis symptoms; antibiotic therapy
MeSH Terms: conditions — Lyme Disease; Lyme Neuroborreliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- definite LNB: patients with definite early Lyme neuroborreliosis
- possible LNB: patients with possible early Lyme neuroborreliosis

SUMMARY:
In this retrospective cohort study of patients with early Lyme neuroborreliosis (LNB), clinical and microbiologic characteristics and long-term outcome of definite vs. possible LNB were evaluated at a single university medical center in Slovenia. Severity of acute disease and long-term outcome during a 12-month follow-up were assessed using a composite clinical score based on objective clinical findings and subjective complaints.

ELIGIBILITY:
Inclusion Criteria:

* early Lyme neuroborreliosis

Exclusion Criteria:

* Not fulfilling study criteria for definite or possible Lyme neuroborreliosis
* Alternative diagnosis during follow-up
* Concomitant tick-borne encephalitis
* Clinical symptoms/signs present for >6 months
* Data not available

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with definite or possible early Lyme neuroborreliosis
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
composite clinical score | follow-up for 12 months-post-treatment
  Composite clinical score based on objective clinical findings and subjective complaints. The sum of subjective complaints and objective findings scored as 0=absent or 1=present represent severity of disease on admission or clinical outcome at follow-up, respectively. Maximum total score=31

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
Only on reasonable request.